CLINICAL TRIAL: NCT05707169
Title: Comparison of Zero- and Two-centimeter Distance From Sapheno-femoral Junction in Laser Ablation of Long Saphenous Vein Incompetence: Evaluating the Kissing Technique
Brief Title: Comparison of Zero- and Two-centimeter Distance From Sapheno-femoral Junction in Laser Ablation of Varicose Vein
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R.22.09.1805 - 2022/09/06
Record Dates: First submitted 2022-09-11; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Varicose Veins; Venous Reflux; Venous Insufficiency; Venous Leg Ulcer
MeSH Terms: conditions — Varicose Veins; Venous Insufficiency; Varicose Ulcer | interventions — Lidocaine; Levobupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Laser Ablation of varicose veins
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two Centimeters from Saphenofemoral Junction (Experimental): Endogenous Laser Ablation (EVLA) uses a laser fibre, which is inserted into the refluxing vein via skin puncture. Using 1470 nm laser and a radial fibre for less discomfort. The catheter is placed 2-2.5 cm distal to the sapheno-femoral junction. Tumescence with a mixture of 20 mL 2% lidocaine, 1: 200,000 adrenaline and 20 mL 0.5% levobupivacaine in 1 L of 0.9% saline
  Interventions: Procedure: Saphenous Ablation; Device: Endogenous Laser Ablation (EVLA); Drug: mixture of 20 mL 2% lidocaine, 1: 200,000 adrenaline and 20 mL 0.5% levobupivacaine in 1 L of 0.9% saline
- Zero point Ablation (Experimental): The catheter is positioned exactly at the terminal valve of the SFJ (kissing the valve).
  Interventions: Procedure: Saphenous Ablation; Device: Endogenous Laser Ablation (EVLA)

INTERVENTIONS:
Procedure: Saphenous Ablation — Endogenous Laser Ablation (EVLA) uses a laser fibre, which is inserted into the refluxing vein via skin puncture.
Device: Endogenous Laser Ablation (EVLA) — Endogenous Laser Ablation (EVLA)
Drug: mixture of 20 mL 2% lidocaine, 1: 200,000 adrenaline and 20 mL 0.5% levobupivacaine in 1 L of 0.9% saline — mixture of 20 mL 2% lidocaine, 1: 200,000 adrenaline and 20 mL 0.5% levobupivacaine in 1 L of 0.9% saline
  Arms: Two Centimeters from Saphenofemoral Junction

SUMMARY:
EVLA is used in in treating refluxing veins, commonly the GSV. The tip of catheter is usually placed 2-2.5 cm distal to the sapheno-femoral junction. This technique theoretically provides the lowest risk for endothermal heat-induced thrombosis (EHIT).

In the present study we aimed to evaluate the zero-distance technique (the kissing technique) compared to 2-cm distance from SFJ valve in ablating incompetent GSV.

DETAILED DESCRIPTION:
INTRODUCTION Chronic venous disease (CVD) is one of the most common pathologies in the general population of adults in both industrialized and developing countries. the most severe form of CVD is venous ulceration with an overall prevalence of about 1 % in the adult population, which increases with age and is more common in women and obese patients. Venous ulcers significantly impair quality of life, and their treatment places a heavy financial burden upon healthcare systems. Varicose veins (VVs) is a common disease in adults, and VVs without skin changes are present in about 20% of the population, while active ulcers are found in 0.5%.The traditional surgical treatment of VVs is high ligation of the great saphenous vein (GSV), axial stripping and phlebotomy, but the postoperative clinical recurrence is as high as 60%.4 Minimally invasive techniques, such as endovenous laser ablation (EVLA) and radiofrequency ablation (RFA), have become widely used for the treatment of VVS. Several reports have shown Several reports have shown that endovenous techniques are as effective as traditional procedures.

EVLA is used in in treating refluxing veins, commonly the GSV. The tip of catheter is usually placed 2-2.5 cm distal to the sapheno-femoral junction. This technique theoretically provides the lowest risk for endothermal heat-induced thrombosis (EHIT).

In the present study we aimed to evaluate the zero-distance technique (the kissing technique) compared to 2-cm distance from SFJ valve in ablating incompetent GSV. Postoperative quality of life (QoL) analysis was assessed using the Aberdeen Varicose Vein Questionnaire (AVVQ) and Venous Clinical Severity Score (VCSS).

Aim of the work: To compare laser therapy ablation of long saphenous vein reflux by conventional and the kissing techniques on development of DVT, recurrence rate of VVs, ulcer-free time, and health-related quality of life.

Patients and methods Study location: The study will be conducted at the department of vascular surgery in Mansoura University, Faculty of Medicine, Mansoura, Egypt .

Type of study: Randomized Controlled Prospective study Study duration: 2 years: 2022-2024 Sample size: It will include all patients presented to our department fulfilling the inclusion criteria.

Study population: The study will be conducted in patients with Incompetent long saphenous vein with and without ulcer.

Inclusion criteria Primary symptomatic VVS (CEAP, C3-C6), sapheno-femoral junction (SFJ) incompetence, and GSV reflux from the groin to below the knee Exclusion criteria included; history of venous surgery, suspected or proven deep venous thrombosis, history of DVT, reflux of deep veins to distal limb, duplication of GSV, and patients' refusal to participate in the trial.

Data collection: The demographics, symptoms, and preoperative clinical data will be collected.

History Data: including underlying medical conditions, any previous associated morbidity.

Examination: Venous examinations. Laboratory: Blood picture, Blood sugar level, Kidney functions, Liver functions and Coagulation profile.

Imaging: Duplex US Method of Randomization: Computer-based Therapies Conventional Technique: Endogenous Laser Ablation (EVLA) uses a laser fibre, which is inserted into the refluxing vein via skin puncture. Using 1470 nm laser and a radial fibre for less discomfort. The catheter is placed 2-2.5 cm distal to the sapheno-femoral junction. Tumescence with a mixture of 20 mL 2% lidocaine, 1: 200,000 adrenaline and 20 mL 0.5% levobupivacaine in 1 L of 0.9% saline.

The kissing technique: The catheter is positioned exactly at the terminal valve of the SFJ (kissing the valve).

Follow up

Criteria for technical success will be:

1. Closed or absent GSV with absent reflux
2. A re-canalized GSV or treatment failure will be defined as an open segment of the treated vein segment of >10 cm in length.
3. All patients are followed in outpatient's settings at 1, 3, 6, 12, and 24 months after surgery.
4. The operation time, number of punctures, intraoperative blood loss (determined by the swabs weighed pre and postoperatively)
5. Recurrence of varicosities and any complications are recorded.

The criteria for assessment:

1. Assessment of Heat induced thrombosis
2. Ecchymosis was confirmed 72 h after operation when the lividity and congestion area was >1 cm2 in the affected limbs.
3. Skin burns were identified 72 h after operation when the skin was red and oedematous according to the criteria for burns.
4. Recurrence was defined by both duplex ultrasound and the clinical examination. A varicose vein that had not been observed before or previously been marked by the patient on the AVVQ form was considered to be a recurrent varicose vein (owing to neo-vascularization or dilation of pre-existing veins).7,11
5. Sensory impairment (numbness) that occurred around incisions was recorded based on the patient's history and physical examination.

QoL assessment The diseased relation effect on QoL was determined using the AVVQ (Chinese version), which assessed the specific effect on QoL and was scored from 0 (no effect of VVS on QoL) to a theoretical maximum of 100.8 The VCSS (Chinese version) was also completed (for the VCSS, 0 represents no significant venous disease and 30 is the maximum score), which is a valid sensitive and responsive measure of the severity of VVs.

Statistical analysis

· The data will be analyzed using Statistical Package for the Social Sciences. The numerical outcomes e.g. age is calculated as mean. Gender will be recorded as frequency and percentage. Chi Square test is applied to assess the association of various parameters. The results will be considered statistically significant if the p-value is found to be less than or equal to 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Primary symptomatic VVS (CEAP, C3-C6), sapheno-femoral junction (SFJ) incompetence, and GSV reflux from the groin to below the knee

Exclusion Criteria:

* history of venous surgery, suspected or proven deep venous thrombosis, history of DVT, reflux of deep veins to distal limb, duplication of GSV, and patients' refusal to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-02-04 (Estimated); Study Completion 2024-05-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 6 months
  both duplex ultrasound and the clinical examination. A varicose vein that had not been observed before or previously been marked by the patient on the AVVQ form was considered to be a recurrent varicose vein (owing to neo-vascularization or dilation of pre-existing veins).

SECONDARY OUTCOMES:
Heat induced thrombosis | 6 months
  Duplex Finding of thrombus near saphenofemoral junction

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rasmussen LH, Bjoern L, Lawaerz M, Lawaetz B, Blemings A, Eklof B. Randomised clinical trial comparing endovenous laser ablation with stripping of the great saphenous vein: clinical outcome and recurrence after 2 years. Eur J Vasc Endovasc Surg 2010;39 — https://pubmed.ncbi.nlm.nih.gov/21725957/
- See also: Subwongcharoen S, Praditphol N, Chitwiset S. Endovenous microwave ablation of varicose veins: in vitro, live swine model, and clinical study. Surg Laparosc Endosc Percutan Tech 2009;19(2):170e4. — https://pubmed.ncbi.nlm.nih.gov/19390287/